CLINICAL TRIAL: NCT05099523
Title: The Effects of Intraoperative Oxygen Used at Different Concentrations on Oxidatıve Stress Markers
Brief Title: Intraoperative Different Concentrations Oxygen And Oxidatıve Stress Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Gamze Küçükosman, Principal investigator, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2021/01
Record Dates: First submitted 2021-09-08; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Stress; Hyperoxia
Keywords: oxidative stress markers; general anesthesia
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Placebo Comparator): 50%Fio2
  Interventions: Procedure: taking arterial blood sample through the injector
- group II (Active Comparator): 30%Fio2
  Interventions: Procedure: taking arterial blood sample through the injector

INTERVENTIONS:
Procedure: taking arterial blood sample through the injector — taking blood samples from patients applied with different oxygen concentrations

SUMMARY:
The aim of the study was to assess the effect of intraoperative oxygen (O2), which was applied at 30% and 50% concentrations on patients who had undergone septoplasty surgery, on Total Oxidant Status (TOS), Total Antioxidant Status (TAS), and Oxidative Stress Index (OSI).

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18-60 years,
* ASA I-II risk class with a minimum operative time of 1.5 hour(s) for whom septoplasty operation under elective conditions

Exclusion Criteria:

* metabolic, endocrine, hepatic, cardiac, or renal diseases,
* malignancies and who used a drug with antioxidant properties such as vitamin E-C
* acetylcysteine in the last 48 hours,
* patients requiring intraoperative 100% O2 inhalation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
EFFECTS OF INTRAOPERATIVE OXYGEN USED AT DIFFERENT CONCENTRATIONS ON OXIDATIVE STRESS MARKERS | end of the surgery
  TAS and TOS values occurring at different oxygen concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes